CLINICAL TRIAL: NCT00170729
Title: Multi-center, Randomized, Double Masked, Vehicle Controlled Phase IV Study to Compare the Efficacy, Ocular Safety and Tolerability of a Two Day Treatment With Eye Drops (0.5% Prednisolone Acetate, One Drop Four Times Per Day) in Patients With Intraocular Inflammation After Cataract Surgery, Followed by an Open Label Observational Period of 12 Days
Brief Title: A Study to Compare Ocular Safety and Tolerability of Eye Drops Containing Prednisolone Acetate in Patients With Intraocular Inflammation After Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ULT 491 A DE 01
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Cataract Surgery
Keywords: Prednisolone acetate,; efficacy,; cataract,; eye drops,; tolerability,; inflammation
MeSH Terms: conditions — Cataract; Inflammation | interventions — prednisolone acetate

INTERVENTIONS:
Drug: Prednisolone acetate

SUMMARY:
The primary objective was to demonstrate that two days of treatment with 0.5% prednisolone acetate eye-drops after cataract surgery are superior to vehicle in reducing the flare in the anterior chamber of the operated eye.

ELIGIBILITY:
Inclusion Criteria:

* Patient gave written informed consent.
* Patient was > 40 years of age.
* Patient had undergone cataract surgery according to standard surgical procedures (see Appendix 2 to the Protocol).
* Patient showed flare in anterior chamber of ≥ 20 photons/msec on Day 1 as compared to the preoperative value measured at screening
* Patient gave written informed consent.

Exclusion Criteria:

* Ophthalmologic conditions
* Operation not performed according to the standard procedures.
* Any eye condition which urgently requires treatment with NSAIDs or corticosteroids.
* History of intraocular surgery in the operated eye.
* Any laser therapy or cryotherapy in the operated eye in the 90 days preceding surgery.
* Any previous episode of uveitis in the operated eye.
* Clinically significant trichiasis or other clinically relevant concurrent inflammatory/ infective eye disorders (e.g. conjunctivitis, episcleritis) except mild forms of seborrheic blepharitis.
* Severe dry eye syndrome.
* Glaucoma.
* Any other clinically significant disorder of the operated eye.
* Contact lens wearer during the treatment period. Systemic conditions
* Hypersensitivity to any of the ingredients of the trial medication.
* Diabetes mellitus (even if currently controlled).
* Severe systemic dysfunction (cardiac, pulmonary, hepatic, renal or endocrine).
* Rheumatoid arthritis.
* Subjects with history of malignancy of any organ system, treated or untreated, within the past five years, whether or not evidence of local recurrence or metastases exists, are excluded, with the exception of localized basal cell carcinoma of the skin.

Prohibited concomitant medication

* Treatment of the eye (to be operated on) with local anti-inflammatory drugs during 14 days preceding surgery and during the trial.
* Systemic use of corticosteroids 4 weeks preceding the surgery and during the trial. Inhaled corticosteroids are allowed if stable 4 weeks preceding the trial and during the trial. Topical corticosteroids to treat dermatological diseases are allowed, too.
* Chronic systemic use of NSAIDs 4 weeks prior to the trial and during the trial, but occasional use (≤ 2 times per week) of NSAIDs or OTC painkillers to treat minor conditions was acceptable. Low dose aspirin for cardiovascular prophylaxis was allowed.

Other prohibited conditions

* Pregnant or lactating women or of childbearing potential unless adequate birth control methods were used throughout the study.
* Mentally handicapped subjects.
* Alcohol/drug abuse.
* Concomitant or recent use of any other investigational agents within 3 months prior to study start.
* Patient's repeated participation in this trial.
* Any medical or laboratory condition which, in the Investigator's opinion, would preclude the participant from adhering to the protocol or completing the trial per protocol.
* participation in another clinical study within 4 weeks prior enrolment;
* have hematological diseases such as aplastic anemia, panmyelopathy, or hemolytic icterus; with severe dysfunction of the liver;
* any medical or laboratory condition which, in the Investigator's opinion, would preclude the participant from adhering to the protocol or completing the trial per protocol;
* subjects with history of malignancy of any organ system, treated or untreated, within the past five years, whether or not evidence of local recurrence or metastases exists, are excluded, with the exception of localized basal cell carcinoma of the skin.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-08-17 (Actual); Primary Completion 2005-02-28 (Actual); Study Completion 2005-02-28 (Actual)

PRIMARY OUTCOMES:
Primary efficacy parameter was the anterior chamber flare of the operated eye, measured by a KOWA laser cell flare meter.

SECONDARY OUTCOMES:
The secondary objectives were to demonstrate that two days treatment with 0.5 % prednisolone acetate eye drops:
are superior to vehicle regarding corneal edema and bulbar conjunctival hyperemia,
are safe regarding intraocular pressure (IOP), visual acuity and frequency of AEs and SAEs,
are well tolerated regarding ocular discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Customer Information, Study Chair — Novartis